CLINICAL TRIAL: NCT01311362
Title: Influence of CYP3A4-induction by St. John's Wort (SJW) on the Steady State Pharmacokinetics of Ambrisentan
Brief Title: Influence of Cytochrome CYP3A4-induction by St. John's Wort on the Steady State Pharmacokinetics of Ambrisentan
Status: Completed | Type: Observational
Sponsor: Gerd Mikus (Other)
Responsible Party: Sponsor-Investigator, Gerd Mikus, Head of Clinical Research Unit, Heidelberg University
Organization: Heidelberg University (Other)
Other Study IDs: K331; 2010-022868-13 (EudraCT Number)
Record Dates: First submitted 2011-03-08; First posted 2011-03-09 (Estimated); Results first posted 2015-06-02 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Drug Interactions
Keywords: Steady-state; Ambrisentan; St. Johns Wort
MeSH Terms: interventions — Hypericum extract LI 160

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- CYP2C19 wild type: CYP2C19 wild type ="extensive metaboliser"
  * Administration of ambrisentan: 5 mg p.o. q.d. on day 1 and days 3-20
  * Administration of St. Johns wort: 300 mg p.o. three times a day (t.i.d.) on days 11-20
  Interventions: Drug: St. Johns wort
- CYP2C19 mutant: CYP2C19 *2/*2 or *2/*3 or *3/*3 = "poor metaboliser"
  * Administration of ambrisentan: 5 mg p.o. q.d. on day 1 and days 3-20
  * Administration of St. Johns wort: 300 mg p.o. three times a day (t.i.d.) on days 11-20
  Interventions: Drug: St. Johns wort

INTERVENTIONS:
Drug: St. Johns wort — * Administration of ambrisentan: 5 mg p.o. q.d. on day 1 and days 3-20
  * Administration of SJW: 300 mg p.o. three times a day (t.i.d.) on days 11-20
  Other Names: Jarsin

SUMMARY:
The aim of the present study is to assess the impact of CYP3A4-induction by SJW on steady state ambrisentan and the impact of the cytochrome P450 2C19 (CYP2C19) genotype (*2 and *3 allele vs. wild type; ~2-5% poor metabolisers in Caucasian population) on the pharmacokinetics of ambrisentan in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Good state of health (physically and mentally)
* Able to communicate well with the investigator, to understand and comply with the requirements of the study
* Voluntarily signed informed consent after full explanation of the study to the participant.
* No clinically relevant findings in any of the investigations of the pre-study examination, especially aminotransferase elevations ≥ 3 × upper limit of normal (ULN). Minor deviations of other laboratory values from normal range may be acceptable, if judged by the investigator to be of no clinical relevance.
* Known genotype for CYP2C19 polymorphism.
* Agreement to abstain from alcoholic beverages during the time of the study.
* Females must agree to use a reliable contraception (Pearl Index <1%), e.g. double barrier method.

Exclusion Criteria:

* Any regular drug treatment within the last two months, except for oral contraceptives in female volunteers and L-thyroxine.
* Any intake of a substance known to induce or inhibit drug metabolising enzymes or drug transporters within a period of less than 10 times the respective elimination half-life or 2 weeks, whatever is longer
* Any participation in a clinical trial within the last month before inclusion
* Any physical disorder which could interfere with the participant's safety during the clinical trial or with the study objectives
* Any acute or chronic illness, or clinically relevant findings in the pre-study examination, especially: a) any condition, which could modify absorption, distribution, metabolism, or excretion of the drug regimen under investigation b) Allergies (except for mild forms of hay fever) or history of hypersensitivity reactions
* Regular smoking
* Blood donation within 6 weeks before first study day
* Excessive alcohol drinking (more than approximately 20 g alcohol per day)
* Inability to communicate well with the investigator due to language problems or poor mental development
* Inability or unwillingness to give written informed consent
* Known or planned pregnancy or breast feeding
* Pre-existing moderate or severe liver impairment
* Contraindication against midazolam, ambrisentan, or SJW or any known intolerance to any of these substances or their additives

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: healthy subjects
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2011-03; Primary Completion 2012-04 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerd Mikus, Prof. Dr., Principal Investigator — deputy head of department
Locations (1):
- University Hospital Heidelberg, Heidelberg, Germany

REFERENCES:
- [Background] Spence R, Mandagere A, Richards DB, Magee MH, Dufton C, Boinpally R. Potential for pharmacokinetic interactions between ambrisentan and cyclosporine. Clin Pharmacol Ther. 2010 Oct;88(4):513-20. doi: 10.1038/clpt.2010.120. Epub 2010 Sep 1. PMID 20811346
- [Background] Harrison B, Magee MH, Mandagere A, Walker G, Dufton C, Henderson LS, Boinpally R. Effects of rifampicin (rifampin) on the pharmacokinetics and safety of ambrisentan in healthy subjects: a single-sequence, open-label study. Clin Drug Investig. 2010;30(12):875-885. doi: 10.2165/11539110-000000000-00000. PMID 20923245

RESULTS

PARTICIPANT FLOW:
Groups:
- Ambrisentan After First Dose: administration of ambrisentan 5 mg p.o. single dose administration of ambrisentan 5 mg p.o. q.d. on day 3-10 administration of ambrisentan 5 mg p.o. q.d on day 11-20 and administration of SJW 300 mg p.o. t.i.d. on day 11-20
Period: Ambrisentan Single Dose
Arm/Group | Ambrisentan After First Dose
Started | 20 (All 20 study participants completed each study period. Total number of study participants: 20)
Completed | 20
Not Completed | 0
Period: Ambrisentan Steady-state
Arm/Group | Ambrisentan After First Dose
Started | 20
Completed | 20
Not Completed | 0
Period: Ambrisentan and SJW
Arm/Group | Ambrisentan After First Dose
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Ambrisentan: administration of ambrisentan 5 mg p.o. single dose administration of ambrisentan 5 mg p.o. q.d. on day 3-10 administration of ambrisentan 5 mg p.o. q.d on day 11-20 and administration of SJW 300 mg p.o. t.i.d. on day 11-20
Arm/Group | Ambrisentan
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.3 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 16
Region of Enrollment [Number; unit: participants]
  Germany | 20

OUTCOME MEASURES:

1. Primary Outcome: AUC of Ambrisentan
Time Frame: after first dose, at steady-state, during St John's wort
Measure: Geometric Mean (95% Confidence Interval); unit: h*ng/ml
Groups:
- Ambrisentan After First Dose: administration of ambrisentan 5 mg p.o. single dose
- Ambrisentan at Steady-state: administration of ambrisentan 5 mg p.o. q.d. on day 3-10
- Ambrisentan During St John's Wort: administration of ambrisentan 5 mg p.o. q.d. on day 11-20 and administration of SJW 300 mg t.i.d. on day 11-20
Arm/Group | Ambrisentan After First Dose | Ambrisentan at Steady-state | Ambrisentan During St John's Wort
Number analyzed (Participants) | 20 | 20 | 20
h*ng/ml | 3670 [3200 to 4220] | 3520 [3120 to 3970] | 2790 [2470 to 3150]

2. Primary Outcome: Cmax of Ambrisentan
Time Frame: after first dose, at steady-state and during St John's wort
Measure: Geometric Mean (95% Confidence Interval); unit: ng/ml
Groups:
- Ambrisentan During St John's Wort: administration of ambrisentan 5 mg p.o. q.d. on day 11-20 and administration of SJW 300 mg p.o. t.i.d. on day 11-20
Arm/Group | Ambrisentan After First Dose | Ambrisentan at Steady-state | Ambrisentan During St John's Wort
Number analyzed (Participants) | 20 | 20 | 20
ng/ml | 447 [397 to 502] | 456 [399 to 521] | 383 [331 to 444]

ADVERSE EVENTS:
Arm/Group | Ambrisentan After First Dose | Ambrisentan at Steady-state | Ambrisentan During St John's Wort
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 14/20 | 14/20 | 6/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ambrisentan After First Dose (N=20) | Ambrisentan at Steady-state (N=20) | Ambrisentan During St John's Wort (N=20)
Headache (General disorders) | 9 | 9 | 4
increase of liver transaminases (Hepatobiliary disorders) | 3 | 3 | 0
nasal congestion (General disorders) | 5 | 5 | 2
Back pain (General disorders) | 1 | 1 | 0
Nasopharyngitis (General disorders) | 1 | 1 | 2
heart palpitation (General disorders) | 1 | 1 | 0
heat sensation (General disorders) | 1 | 1 | 0
thoracic discomfort (General disorders) | 1 | 1 | 0
flush (General disorders) | 1 | 1 | 0
pressure sensation in head (General disorders) | 1 | 1 | 1
diarrhoea (General disorders) | 1 | 1 | 0
nightmares (General disorders) | 1 | 1 | 0

LIMITATIONS AND CAVEATS:
The extent of this interaction was small and thus likely without clinical relevance.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No